CLINICAL TRIAL: NCT06117241
Title: A Transdisciplinary Approach to Investigating Metabolic and Risk of Early-Onset Colorectal Cancer: A Randomized Intervention Trial in Human Dyads and Mechanistic Study in Animals
Brief Title: Reducing Metabolic Dysregulation in Dyads
Acronym: REMEDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, James Hebert, Health Sciences Distinguished Professor; Director, Cancer Prevention and Control Program, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00120270
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Inflammation; Nutrition Related Cancer
Keywords: Body Composition; Cancer; Digestive System; Microbiome
MeSH Terms: conditions — Colorectal Neoplasms; Inflammation; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison (No Intervention): Participation will be for six months. Participants will meet staff at three timepoints (baseline, 3 months, 6 months) to complete questionnaires, online dietary assessment, body measures, have blood pressure measured, provide blood and stool samples, and wear an activity monitor for a week at each time point.
- Intervention (Experimental): Participation will be for six months. Participants will meet staff at three timepoints (baseline, 3 months, 6 months) to complete questionnaires, online dietary assessment, body measures, have blood pressure measured, provide blood and stool samples, and wear an activity monitor for a week at each time point. In addition, participants will attend weekly classes for 12 weeks and one class per month for three months. These classes will include cooking, movement, and stress reduction.
  Interventions: Behavioral: IMAGINE HEALTHY

INTERVENTIONS:
Behavioral: IMAGINE HEALTHY — An anti-inflammatory nutrition program including cooking classes, physical activity, and stress reduction.
  Arms: Intervention

SUMMARY:
This study is a 6-month randomized controlled trail of diet modification designed to reduce chronic inflammation and reverse metabolic dysfunction among obese individuals with one or more polyps found at a colonoscopy screening. We also will recruit an at least overweight partner, who lives in the same household. To be eligible, participants will be apparently disease-free, obese AAs or EAs who have self-identified a partner who is at least 9 years, with whom they live and who also is at least overweight. Each index participant will: 1) Be AA or EA by self-report; 2) Be ≤55 years old; 3) Have undergone a colonoscopy screening and found to have ≥1 polyp(s); 4) Be free of co-morbid conditions or other factors that would limit participation in this trial; 5) Have a BMI ≥30kg/m2; 6) Be willing to commit to investing the time and effort required to participate in this trial (i.e., willing to complete all assessments and provide biological samples as specified in the consent); and 7) Have no recent antibiotic use. Their partner needs to: 1) Be at least 9 years old; 2) Live in the same household and consumes meals together; 3) Be at least overweight; 4) Agree to all study procedures, including provision of biological samples, body measurements, and self-reported dietary and other assessments; and 5) Have no recent antibiotic use.

DETAILED DESCRIPTION:
This project leverages our expertise in the epidemiology of colorectal cancer (CRC); disparities; obesity; metabolic dysregulation, an important manifestation of inflammation; the microbiome; animal CRC models; and lifestyle intervention trials to address the growing problem of Early-Onset CRC (EOCRC) (i.e., <50 years). Adiposity and diet drive metabolic dysregulation. So, understanding the interaction between diet and adiposity are key to understanding the genesis of EOCRC - and an array of other obesity-related cancers. This project will address the absence of critical clinical trials and mechanistic studies involving lifestyle interventions for EOCRC. We intend to address this gap; and have the transdisciplinary team representing complementary backgrounds to do so. We focus on dietary modulation of gut microbes to reduce metaflammation and subsequent metabolic dysfunction in obesity, with a goal of preventing EOCRC. We will perform an anti-inflammatory dietary intervention trial in dyads of adults and children at elevated risk for CRC. We also will conduct a complementary mechanistic animal study that builds on and leverages our expertise in mechanistic studies on obesity and CRC. This work is supported by infrastructure that we have built over the past decades in two key centers at the University of South Carolina (USC): (1) Center for Colon Cancer Research (CCCR, 2002 - present - which specializes in mouse models of CRC); and (2) the Cancer Prevention and Control Program (CPCP, 2003 - present - which specializes in the epidemiology of cancer and lifestyle intervention trials for cancer, with a focus on cancer disparities). The two projects that comprise the proposed grant address two Specific Aims that are represented by the human study and laboratory animal experiment: i.e. ,1: To establish the metabolic protective effects of an anti-inflammatory diet in obese, high-risk African-American (AA) and European-American (EA) adults and children in reducing inflammation as indicated by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), IGF-1, Tumor Necrosis Factor alpha (TNFα), Interleukin 6 (IL-6), and C-Reactive Protein (CRP), and a creating more favorable microbiome signature; 2: To establish gut microbes as mediators between anti-inflammatory dietary input and reversal of metabolic dysfunction and associated CRC risk. This complements the human study by carrying out pre-clinical murine model studies with similar inputs (diet), intermediate endpoints (inflammation, microbiome), and outcomes (CRC-related). We hypothesize that an anti-inflammatory dietary intervention will reduce metabolic dysfunction and metainflammation through regulatory effects on gut microbiota.

Results from this work will address the role of metabolic dysregulation in relation to factors that are known to be important in carcinogenesis, that therefore could have profound effects on EOCRC, have implications for other obesity-related cancers, and have great promise for moving the field forward by addressing mechanisms that drive large health-related disparities that consistently disfavor African Americans.

ELIGIBILITY:
Individuals eligible to participate in this study will be apparently disease- free, obese (BMI ≥ 30kg/m2) AAs or EAs who have self-identified a partner who is at least 9 years old, with whom they live and who also is at least overweight. Each index patient will: 1) Be AA or EA by self-report; 2) Be ≤55 years old; 3) Have agreed to undergo colonoscopy screening and found to have ≥1 polyp(s) that place them at elevated risk for future adenomas and CRC; 4) Be free of co-morbid conditions or other factors that would limit participation in this trial; 5) Have a BMI ≥30kg/m2; 6) Be willing to commit to investing the time and effort required to participate in this trial (i.e., willing to complete all assessments and provide biological samples as specified in the consent); and 7) Have no recent antibiotic use (≤3 months). Their dyad partner needs to: 1) Be at least 9 years old; 2) Live in the same household and consumes meals together; 3) Be at least overweight; 4) Agree to all study procedures, including provision of biological samples, anthropometric measurements, and self-reported dietary and other assessments; 5) Have no recent antibiotic use (≤3 months).

Ages: 9 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood | Baseline, 3-month, 6-month
  Tumor Necrosis Factor alpha (TNFα), Interleukin 6 (IL-6), and C-Reactive Protein (CRP)
Stool | Baseline, 3-month, 6-month
  Determine race-specific microbiome signatures associated with anti-inflammatory dietary input and reversal of metabolic dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The information collected for this study will also be transferred into a secure, electronic database at the Biostatistics Center of George Washington University. The database will have information from all the participants as well as from other related studies. Information will not include directly identifying information such as name, address, social security number, or medical record number. The study will use a unique code for each person consisting of a set of letters and numbers. The key to the code linking the data to the participant will be kept at USC in a secure manner. Information in the database will only be used for statistical analyses. At the conclusion of the study, some biological samples as well as data from USC may be shared with biospecimen and data repositories supported by the NIH, which funded this study. Data and biological samples sent to these repositories will be identified only by a code number and cannot be linked to a participant.
Supporting Information: Study Protocol, SAP